CLINICAL TRIAL: NCT07019610
Title: Evaluation of Chlorhexidine Caps for Central Line Associated Blood Stream Infection Prevention in People Needing Hemodialysis: a Pilot Randomised Control Trial
Brief Title: Chlorhexidine Caps for CLABSI Prevention in Hemodialysis: a Pilot Randomized Controlled Trial
Acronym: ECHO-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IVPA_25.01
Record Dates: First submitted 2025-06-02; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Vascular Access Complication; Device Related Infection; Device Related Sepsis; Catheter Infection; Catheter Complications; Catheter-Related Infections; Catheter Related Complications; Hemodialysis Catheter Infection; Hemodialysis Catheter-associated Infection; Hemodialysis Complication
Keywords: Hemodialysis Catheter; Randomised Controlled Trial; Antimicrobial Barrier Caps; Vascular access device; Hemodialysis catheter caps; Chlorhexidine cap; Central Venous Catheter; CVC; CLABSI; Central Line Associated Blood Stream Infection
MeSH Terms: conditions — Prosthesis-Related Infections; Catheter-Related Infections

STUDY DESIGN:
Intervention Model Description: A single-centre, two-arm, parallel group randomised controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Standard Non-Antimicrobial Hemodialysis Cap
  Interventions: Device: B Braun Combi-stopper
- Intervention (Experimental): Antimicrobial Haemodialysis Catheter Luer End Cap
  Interventions: Device: ClearGuard HD

INTERVENTIONS:
Device: ClearGuard HD — The ClearGuard HD end cap is a male luer lock end cap that incorporates an antimicrobial treatment (Chlorhexidine) on its surface designed to reduce microbial colonisation within a haemodialysis catheter hub.
  Other Names: Haemodialysis Catheter Luer End Cap
  Arms: Intervention
Device: B Braun Combi-stopper — Standard practice caps used within the Metro North Kidney Health Service
  Other Names: Standard Non-Antimicrobial Hemodialysis Cap
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare a chlorhexidine antimicrobial barrier cap in patients requiring hemodialysis treatment to the standard hemodialysis caps currently used within the Metro North Kidney Health Service.

The main questions to answer are:

* Study Feasibility
* Occurrence of infectious complications related to renal central venous catheters

Participants will be randomly allocated to receive either of the below hemodialysis caps to cover their hemodialysis catheter hub:

* The standard hemodialysis cap used at the Royal Brisbane and Women's Hospital, or
* The intervention hemodialysis cap containing chlorhexidine inside it

Researchers will compare standard and chlorhexidine hemodialysis caps to see if the presence of chlorhexidine improves the occurrance of infectious complications related to the hemodialysis catheter.

DETAILED DESCRIPTION:
This study is a single-centre, two-arm, parallel group Randomized Controlled Trial (RCT) to test the effectiveness, safety, impact of device application on health-related quality of life measures, and cost-effectiveness of ClearGuard™ HD antimicrobial barrier caps in patients receiving hemodialysis.

Setting and Sample:

The ECHO-HD will be undertaken at the Metro North Kidney Health Service (MNKHS), Royal Brisbane and Women's Hospital in Queensland, Australia.

Sample Size:

The investigators will recruit 60 patients with 30 patients per arm. The purpose of the pilot study is to assess research project feasibility and inform the design of a large scale powered RCT. Viechtbauer et al. (2015) determined that a sample size of 59 participants is sufficient to detect a problem with a 5% probability of occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Able to provide informed consent
* Kidney failure requiring a tunnelled CVC for treatment (haemodialysis)
* 21 days BSI free
* No known allergy to chlorhexidine and/or nylon and/or polypropylene.

Exclusion Criteria:

* Current CLABSI
* Known allergic to chlorhexidine and/or nylon and/or polypropylene.
* Patients on an end-of-life pathway
* People with a cognitive impairment and/or intellectual disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Eligibility | 12 Months
  Study Eligibility as per inclusion/exclusion criteria (≥80% of screened participants will be eligible for study inclusion)
Recruitment | 12 Months
  Participant Recruitment onto study (≥80% of eligible participants will provide informed consent to participate in the study)
Fidelity | 12 Months
  Protocol fidelity of study participants (≥80% will receive the allocated intervention)
Missing data | 12 Months
  Missing data for primary outcome (<5% of primary outcome data will be unable to be collected).

SECONDARY OUTCOMES:
Central Line Associated Blood Stream Infection (CLABSI) Rates | 12 months with 3 month follow up
  CLABSIs incidence rates (reported as the CLABSI rate per 1000 central line days, which is calculated by dividing the number of CLABSIs by the number of central line days and multiplying the result by 1000 (CDC, 2024)
  Hospitalisation days for CLABSI
Catheter Related Infections | 12 months with 3 month follow up
  Central line related infections, defined as infections other than bloodstream infections caused by a central line insertion/insitu such as local skin infections etc.
Central Venous Catheter (CVC) Failure | 12 months with 3 month follow up
  Central Venous Catheter (CVC) failure/complications (catheter removal due to infection, occlusion and other complications)
Antibiotic Use | 12 months with 3 month follow up
  Antibiotic use (starts due to CLABSI, duration)
Health-related quality of life scores | 12 months with 3 month follow up
  Health-related quality of life scores using EuroQual 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire (see attached User Agreement and EQ-5D-5L Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claire Rickard, Principal Investigator — The University of Queensland
Locations (1):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No